CLINICAL TRIAL: NCT03282175
Title: Effects of Elastic Resistance Training on Physical Performance, Inflammatory Marker and Myokines in Elderly Women
Brief Title: Effects of Elastic Resistance Training on Performance and Biochemical Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UP-FVZ-ERT-Myokine
Record Dates: First submitted 2017-09-06; First posted 2017-09-13 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Exercise
Keywords: BDNF; interleukin-15; interleukin-8; resistin; SPPB
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): Participant in this group performed an acute resistance exercise protocol. The exercise protocol consisted of general warm-up of 10 min, followed by 8 exercises with 2 sets of 8 repetition and 1 min between sets.
  Interventions: Other: Exercise
- Training (Experimental): Participants allocated to intervention group initiated the progressive resistance training program of moderate intensity, with three weekly sessions throughout the 12-week treatment period.
  Interventions: Other: Training
- Control group (Active Comparator): Participants allocated to control group did not receive any placebo or treatment.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Exercise — Exercise session consisted of general warm-up of 10 min, followed by 35-40 min of resistance exercises (chair squats, band seated: biceps curl, seated row, knee extension, leg press and hip abduction; standing behind the chair: knee flexion, and calf rise), and general cool down of 10 min.
  Arms: Exercise
Other: Training — Each training session consisted of general warm-up of 10 min, followed by 35-40 min of resistance exercises (chair squats, band seated: biceps curl, seated row, knee extension, leg press and hip abduction; standing behind the chair: knee flexion, and calf rise), and general cool down of 10 min.
  Arms: Training
Other: Control group — The control group did not receive any treatment.
  Arms: Control group

SUMMARY:
The aim of this study was to investigate the acute and chronic effect of elastic resistance exercise in elderly women living in a nursing home. The primary outcome was the functional performance and hand grip strength. The secondary outcomes were myokines and inflammatory markers analysis.

DETAILED DESCRIPTION:
Evidence regarding the relationship between RT and systemic myokine responses, as well as inflammation and physical performance in elderly is limited. Thus, this study aimed to evaluate the effect of short-term progressive elastic resistance training on muscular strength and physical performance, as well as the acute and chronic response of myokines and inflammatory markers after resistance exercise in elderly women living in a nursing home. From January to February 2016, we invited 95 older women (≥ 65 years) living in nursing home in the south of Slovenia to participate in our study.

The experimental design consisted of 1) baseline testing; 2) acute elastic resistance exercises with post-exercise and 2h post-exercise biochemical analysis; 3) a 3 months of supervised, progressive elastic resistance training program of moderate intensity; and 4) post-training testing.

The quantification of biomarkers was done using the MAGPIX® system, magnetic bead-based multi-analyte panels and MILLIPLEX® Analyst 5.1 software (MAGPIX®, Merck Millipore) and a human premixed 4-plex kit (R&D System Inc., Minneapolis, MN, USA), strictly following the manufacturer's instructions.

Two-way mixed ANOVA model was used to test group × time interaction. Tukey's post hoc test was applied for statistically significant interaction. To test for significant differences between groups relating anthropometric and biochemical variables, we used a Student's t-test. All values are expressed as mean and standard deviation (SD). P values of <0.05 is considered statistically significant. Bonferroni's correction for multiple testing will be performed by multiplying the P value with the number of tests where appropriate. Statistical analyses will be carried out using the SPSS program, version 21 (Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* nursing home residents
* participants did not perform any regular resistance training

Exclusion Criteria:

* immobility
* implantable cardiac peacemaker
* severe dementia
* terminal illness

Ages: 65 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Female nursing home residents
Enrollment: 20 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Functional performance | 1 week
  A short battery of physical performance tests (SPPB) was used to assess baseline and post-training lower extremity function (0-12 point scale).

SECONDARY OUTCOMES:
Acute effect of resistance exercise | 4 hours
  The acute effect of resistance exercise on plasma concentrations of myokines and inflammatory markers measured pre-, post- and 2h post-exercise.
Biochemical analysis of chronic effect of resistance training | 2 weeks
  The chronic effect of resistance training on plasma concentrations of myokines and inflammatory markers measured at baseline and post-training.

CONTACTS AND LOCATIONS:
Overall Officials: Felicita Urzi, MSc, Principal Investigator — University of Primorska Faculty of Mathematics, Natural Sciences and Information Technologies

REFERENCES:
- [Background] Argiles JM, Lopez-Soriano FJ, Busquets S. Therapeutic potential of interleukin-15: a myokine involved in muscle wasting and adiposity. Drug Discov Today. 2009 Feb;14(3-4):208-13. doi: 10.1016/j.drudis.2008.10.010. Epub 2008 Dec 16. PMID 19041416
- [Background] Busquets S, Figueras M, Almendro V, Lopez-Soriano FJ, Argiles JM. Interleukin-15 increases glucose uptake in skeletal muscle. An antidiabetogenic effect of the cytokine. Biochim Biophys Acta. 2006 Nov;1760(11):1613-7. doi: 10.1016/j.bbagen.2006.09.001. Epub 2006 Sep 12. PMID 17056184
- [Background] Geroldi D, Minoretti P, Emanuele E. Brain-derived neurotrophic factor and the metabolic syndrome: more than just a hypothesis. Med Hypotheses. 2006;67(1):195-6. doi: 10.1016/j.mehy.2006.02.001. Epub 2006 Mar 20. No abstract available. PMID 16545915
- [Background] Martins WR, Safons MP, Bottaro M, Blasczyk JC, Diniz LR, Fonseca RM, Bonini-Rocha AC, de Oliveira RJ. Effects of short term elastic resistance training on muscle mass and strength in untrained older adults: a randomized clinical trial. BMC Geriatr. 2015 Aug 12;15:99. doi: 10.1186/s12877-015-0101-5. PMID 26265075
- [Background] Oesen S, Halper B, Hofmann M, Jandrasits W, Franzke B, Strasser EM, Graf A, Tschan H, Bachl N, Quittan M, Wagner KH, Wessner B. Effects of elastic band resistance training and nutritional supplementation on physical performance of institutionalised elderly--A randomized controlled trial. Exp Gerontol. 2015 Dec;72:99-108. doi: 10.1016/j.exger.2015.08.013. Epub 2015 Sep 2. PMID 26341720
- [Background] Prestes J, Shiguemoto G, Botero JP, Frollini A, Dias R, Leite R, Pereira G, Magosso R, Baldissera V, Cavaglieri C, Perez S. Effects of resistance training on resistin, leptin, cytokines, and muscle force in elderly post-menopausal women. J Sports Sci. 2009 Dec;27(14):1607-15. doi: 10.1080/02640410903352923. PMID 19967592
- [Background] Pereira DS, de Queiroz BZ, Miranda AS, Rocha NP, Felicio DC, Mateo EC, Favero M, Coelho FM, Jesus-Moraleida F, Gomes Pereira DA, Teixeira AL, Maximo Pereira LS. Effects of physical exercise on plasma levels of brain-derived neurotrophic factor and depressive symptoms in elderly women--a randomized clinical trial. Arch Phys Med Rehabil. 2013 Aug;94(8):1443-50. doi: 10.1016/j.apmr.2013.03.029. Epub 2013 Apr 18. PMID 23602881
- [Background] Troseid M, Lappegard KT, Claudi T, Damas JK, Morkrid L, Brendberg R, Mollnes TE. Exercise reduces plasma levels of the chemokines MCP-1 and IL-8 in subjects with the metabolic syndrome. Eur Heart J. 2004 Feb;25(4):349-55. doi: 10.1016/j.ehj.2003.12.006. PMID 14984925
- [Background] Yeo NH, Woo J, Shin KO, Park JY, Kang S. The effects of different exercise intensity on myokine and angiogenesis factors. J Sports Med Phys Fitness. 2012 Aug;52(4):448-54. PMID 22828466